CLINICAL TRIAL: NCT05371990
Title: A Cross-sectional Study on the Evaluation of Nutritional Habits of Students at Istanbul Medeniyet University.
Brief Title: Evaluation of Nutritional Habits of University Students
Status: Completed | Type: Observational
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Gülin Öztürk Özkan, Head of department (PhD) Assistant Professor, Istanbul Medeniyet University
Other Study IDs: 2020/39
Record Dates: First submitted 2022-05-05; First posted 2022-05-12 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2022-05

CONDITIONS: Eating Habit; Health Knowledge, Attitudes, Practice
MeSH Terms: conditions — Feeding Behavior; Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Determination of Eating habits — Questionnaire

SUMMARY:
This cross- sectional, single-center study was conducted with the participation of 912 students studying at [removed for blind peer review] Faculty of Health Sciences, Faculty of Engineering and Natural Sciences, Faculty of Educational Sciences, Faculty of Social Sciences, Faculty of Law and Medicine. The sample size was calculated to be a minimum of 379 with 95% confidence over the total number of students, 5301. The study was carried out between October 2020 and December 2020. The compliance of the study with the ethical rules was evaluated by the Istanbul Medeniyet University Social and Human Sciences Research and Publication Ethics Committee at its meeting dated 27.10.2020 and approved with the decision numbered 2020/39.

At the beginning of the study, verbal and written consent was obtained from the individuals and a questionnaire containing 29 questions was distributed by the researchers. The questionnaire form consists of three parts. The first part includes 10 questions to determine the demographic characteristics of the participants, the second part includes 17 questions to determine their eating habits, and the third part includes 2 questions to evaluate the status of following the news about nutrition and heart health and whether they find the public service ads on this subject sufficient.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the research
* Istanbul Medeniyet University students between the ages of 18-25

Exclusion Criteria:

* Individuals who did not volunteer to participate in the study
* Adults over 25
* All university students studying outside of Istanbul Medeniyet University
* Elderly individuals
* Children under 18

Ages: 18 Years to 25 Years | Sex: All
Age Groups: Adult
Study Population: University students studying at Istanbul Medeniyet University and volunteering to participate in the research
Sampling Method: Probability Sample
Enrollment: 912 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Reaching the targeted participant | One month
  Participants will be surveyed and evaluated with data obtained using appropriate statistical methods.

CONTACTS AND LOCATIONS:
Locations (1):
- İstanbul Medeniyet University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No